CLINICAL TRIAL: NCT05166720
Title: Clinical Application of the Best Evidence of NIDCAP in Very Low Birth Weight Infants
Brief Title: Application of the Best Evidence of Neonatal Individualized Developmental Care Assessment Program (NIDCAP) in Very Low Birth Weight Infant (VLBWI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Huxiaojing
Record Dates: First submitted 2021-10-24; First posted 2021-12-22 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: NIDCAP

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIDCAP care (Experimental): The training core group was formed by the project team. After a one-month clinical unified training on the best evidence of NIDCAP for the VLBW nursing professional group, the best evidence of NIDCAP was applied to the intervention group.
  Interventions: Behavioral: NIDCAP care
- routine nursing care (No Intervention): routine nursingPerform routine care for NICU infants according to the nursing routine of each hospital

INTERVENTIONS:
Behavioral: NIDCAP care — NIDCAP care was performed according to the best evidence of NIDCAP
  Arms: NIDCAP care

SUMMARY:
In order to help THE GROWTH and development of VLBWI in Neonatal Intensive Care Unit (NICU) and reduce the interference of external environment to them, we summarized the best evidence of NIDCAP care, and applied the evidence to the intervention group, and observed the compliance of nurses in the intervention group to the application of evidence, and the short-term outcomes of VLBWI.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1500g;
* admit within 24 hours of birth;
* The guardian signs the informed consent;
* OI (oxygenation index >300)

Exclusion Criteria:

* Newborn with severe congenital malformations or various chromosomal diseases, genetic metabolic diseases, severe neurological diseases;
* Newborn who did not achieved discharge or death at the end of the study period

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Mean length of stay of VLBWI | From the day the VLBWI admitted to the day VLBWI discharged, about two months.
  The average length of stay of VLBWI in the intervention group minus the average length of stay of VLBWI in the control group

SECONDARY OUTCOMES:
Nurse compliance with NIDCAP evidence content | From the beginning of the NIDCAP intervention to the end of the NIDCAP intervention, about three months.
  Members of the study core team will regularly check the NICU nurse's performance by using the checklist. The number of times the NICU nurse performed specified operations divided by the total number of inspections. The checklist includes: Whether bed units and equipments are placed in accordance with the requirements? Whether sound is controlled in the NICU? Whether the skin of VLBWI is taking good care of, etc. Points are awarded if the requirements are met. Higher scores indicate better nurse compliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Research Group of Developmental Care for Very Low Birth Weight Infants in China; Lyu T, Ye R, Li LL, Zhang LL, Xiao J, Ma YL, Li F, Rong H, Liu D, Wang H, Wang Y, Gu WW, Xuan Y, Chen X, Fan QL, Tang YF, Huang XH, Qin A, Zhang YL, Dou Y, Hu XJ. The effect of developmental care on the length of hospital stay and family centered care practice for very low birth weight infants in neonatal intensive care units: A cluster randomized controlled trial. Int J Nurs Stud. 2024 Aug;156:104784. doi: 10.1016/j.ijnurstu.2024.104784. Epub 2024 May 5. PMID 38788261